CLINICAL TRIAL: NCT06801717
Title: Split-Face Comparison of 532nm Potassium Titanyl Phosphate (KTP) Laser Treatment Versus Radiofrequency Microneedling in Combination With 532 KTP Laser for Erythematotelangiectatic or Papulopustular Rosacea
Brief Title: Rosacea Radiofrequency Microneedling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: CynosureLutronic (Industry)
Responsible Party: Principal Investigator, Ariel Eva Eber, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240859
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-01

CONDITIONS: Rosacea, Papulopustular; Rosacea, Erythematotelangiectatic
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Potassium titanyl phosphate (KTP) Laser Therapy with unilateral Radiofrequency Microneedling (Experimental): Participants will be in this group for up to 36 weeks
  Interventions: Device: KTP Laser Therapy; Device: Radiofrequency microneedling

INTERVENTIONS:
Device: KTP Laser Therapy — Participants will receive full face treatments with 532 nm KTP laser for 3 sessions at 8-12 weeks apart. Laser therapy will be conducted in person. Each laser treatment session will last up to 10 minutes.
Device: Radiofrequency microneedling — Participants will receive unilateral facial treatments with radiofrequency microneedling device for 3 sessions at 8-12 weeks apart. Radiofrequency microneedling will be conducted in person. Each treatment session will last up to 1 hour.

SUMMARY:
There are 3 main objectives of this proposal as follows: (1) to assess the efficacy of radiofrequency microneedling in the treatment of erythematotelangiectatic and or papulopustular rosacea, (2) to determine the potential for combination treatment of radiofrequency microneedling with the 532 nm KTP laser, and (3) identify potential novel therapeutic strategies for the treatment of rosacea.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult (>18yo) subjects in general good health
2. Clinical and/or histologic diagnosis of erythematotelangiectatic or papulopustular rosacea.
3. Subject is able to understand and sign informed consent
4. Subject is able to complete the study and comply with study procedures

Exclusion Criteria:

1. Patients currently utilizing oxymetazoline or brimonidine.
2. Presence of dermatoses that might interfere with diagnosis as determined by a study investigator
3. Presence of extreme light sensitivity, or conditions pre-disposing to light sensitivity such as but not limited to xeroderma pigmentosum
4. Any significant medical condition that may prevent the patient from participating in the study according to the investigator's assessment
5. History of poor wound healing or blood-clotting abnormality
6. History of keloid formation or hypertrophic scarring
7. Hypersensitivity or contraindication to local anesthetics as determined by the principal investigator or other medical professional.
8. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Rosacea severity measured by the Clinician's Erythema Assessment (CEA) | Baseline, up to 16 weeks after the last treatment
  Score range from 0 (clear skin) to 4 (severe erythema). Lower scores indicate less rosacea severity as assessed by the CEA scale.

SECONDARY OUTCOMES:
Change in Patient reported impact on quality of life (QOL) measured by DLQI | Baseline, up to 16 weeks after the last treatment
  Dermatology Quality of Life Index (DLQI) is a validated 10-item questionnaire assessing the impact of dermatological conditions on a patient's QOL, with scores ranging from 0 (no impact) to 30 (extremely large impact). Higher scores indicate higher impact on QOL.
Change in patient satisfaction with treatment outcomes measured by Patient Self-Assessment (PSA) | Baseline, up to 16 weeks after the last treatment
  The PSA scale measures the patient's subjective satisfaction with skin's appearance on a scale of 0 (clear of unwanted redness) to 4 (completely unacceptable redness). Higher scores indicate less satisfaction.
Change in Global Aesthetic Improvement scale (GAIS) | Baseline, up to 16 weeks after the last treatment
  The GAIS scores range from 1 (very much improved) to 5 (the appearance is worse than the original condition). Higher scores indicate less satisfaction.
Proportion of blinded photo assessment | Baseline, up to 16 weeks after the last treatment
  Proportion of identification of before and after photos by three blinded rosacea experts will be reported. Expert identification greater than or equal to 80% or greater will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Eber, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Dermatology Miami Beach Clinic, Miami Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No